CLINICAL TRIAL: NCT04060927
Title: LCI-LUN-SBRT-002: Pilot Study of SGRT Alone vs. SGRT in Combination With Fiducials for Breath Hold SBRT Treatments of the Lung
Brief Title: Pilot Study of SGRT Alone vs. SGRT With Fiducials for Breath Hold SBRT tx of the Lung
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081383; 00036616 (Other: Advarra IRB); LCI-LUN-SBRT-002 (Other: Atrium)
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: NSCLC; Lung; Radiation Therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1 (Experimental): Freebreathing SBRT with SGRT
  Interventions: Device: SGRT
- Group 2 (Experimental): Breath hold SBRT with SGRT
  Interventions: Device: SGRT
- Group 3 (Experimental): Breath hold SBRT with SGRT in combination with implanted fiducials
  Interventions: Device: SGRT

INTERVENTIONS:
Device: SGRT — Surface Guided Radiation Therapy

SUMMARY:
This is a pilot study designed to to provide data and experience comparing two different techniques of breath hold SBRT treatments. The first technique will include SGRT, but with the assistance of implanted fiducials. Subjects will be treated with a breath hold technique utilizing SGRT, but will also be imaged during treatment with fiducial match. The second technique will utilize SGRT for breath hold treatments without the assistance of implanted fiducials/continuous imaging.

DETAILED DESCRIPTION:
The study's primary objective is estimate the incidence of SBRT and fiducial-related pulmonary toxicities for subjects treated with SBRT who have tumors that move ≥ 1 cm in 3 different cohorts: 1) free breathing with SGRT 2) breath hold utilizing SGRT only; 3) breath hold utilizing SGRT in combination with implanted fiducials. Secondary objectives also include Estimate reliability of gated SBRT treatments utilizing SGRT vs. SGRT with fiducials estimating local control for SBRT in subjects treated in the three different cohorts, estimating overall survival, and evaluating quality of life. A safety objective of estimating acute and long-term grade 2 or higher non-hematologic toxicities attributed to SBRT/fiducial implantation in subjects treated in the three different cohorts will also be explored.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent with HIPAA authorization for release of personal health information.
2. Age ≥18 years at the time of consent. Because no dosing or adverse event data are currently available on the use of fiducials in combination with SBRT in subjects <18 years of age, children are excluded from this study.
3. ECOG Performance Status of ≤ 2.
4. Stage IA-IIB (T1a-T3bN0) presumed non-small cell lung cancer, carcinoid tumors, or lung metastasis that have ≥ 1 cm of respiratory associated motion measured on 4DCT at time of simulation for SBRT with or without respiratory motion suppression techniques. Histologic confirmation of malignancy is encouraged but not required. Primary or metastatic tumor ≤ 7 cm.
5. Subjects may be receiving systemic chemotherapy or other systemic agents prior to enrollment, but these agents must be stopped during SBRT treatments.
6. Females of childbearing potential (FCBP) must have a negative serum pregnancy test within 14 days prior to day 1 of treatment. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause).
7. The effects of radiation on the developing human fetus are not well described. For this reason, women of child-bearing potential and non-sterilized men who are sexually active with a woman of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. FCBP must be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) from the time of informed consent until 5 days after last dose of SBRT. Contraceptive methods with low user dependency are preferable but not required.
8. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

1. Prior radiation to the chest that would overlap with the current radiation fields and determined by the treating physician to impede the treatment of the study malignancy.
2. Active ongoing pulmonary infection or pneumonitis that is requiring active treatment with antibiotics or steroids. Prior pneumonitis from drug or other therapies that has been treated within 15 days of first day of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of SBRT and fiducial-related pulmonary toxicities as assessed by NCI CTCAE v.5.0 | 12 months
  The outcome will be recorded as a binary variable determined for each subject indicating whether or not the subject had at least one grade 2 or higher pulmonary toxicity related to SBRT or implantation of fiducials.

SECONDARY OUTCOMES:
Reliability of gated SBRT treatments utilizing SGRT vs. SGRT with fiducials | approx. 2 weeks
  This will be recorded as numerical values for each of the shift/rotational directions and the vector composites of the directional shifts at the time of verification imaging.
Local control of treated tumor(s) | up to 24 months
  The outcome will be measured as the duration of time from enrollment to progression of the subject's treated tumor(s)
Overall Survival | approx. 5 years
  This outcome will be measured as the duration of time from the date of enrollment to the study to the date of death from any cause.
Change from Baseline in MD Anderson Symptom Inventory - Lung Cancer (MDASI-LC) Score | pre-SBRT and 1, 3, 6, and 12 months after the last treatment of SBRT
  The MDASI-LC Module includes 22 questions to assess the severity of multiple lung cancer-related symptoms and the impact of these symptoms on daily functioning. Scores for each item range from 0 to 10, where 0 indicates no symptoms and 10 indicates worst possible symptoms.

OTHER OUTCOMES:
Incidence of Grade 2 or higher non-hematologic toxicities attributed to SBRT and fiducial implantation | up to 12 months after the last treatment of SBRT
  Incidence rates for acute and long-term adverse events of special interest, SAEs, and deaths from the time of initiation of SBRT until 12 months after the last treatment of SBRT will be summarized as counts and proportions.

CONTACTS AND LOCATIONS:
Overall Officials: John Heinzerling, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT04060927/ICF_000.pdf